CLINICAL TRIAL: NCT03638050
Title: The Safety of the 6-minute Walk Test After Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Solange Guizilini, Principal Investigator, Federal University of São Paulo
Other Study IDs: 58277816.7.0000.5505
Record Dates: First submitted 2018-07-27; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Acute Myocardial Infarction; Six-minute Walk Test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- In-hospital acute myocardial infarction patients: Functional Capacity Assessment
  Interventions: Other: Functional Capacity Assessment

INTERVENTIONS:
Other: Functional Capacity Assessment — Individuals will be assessed on the third day after acute myocardial infarction. The six-minute walk test will be performed according to the norms of the American Thoracic Society.

SUMMARY:
Background: The six-minute walk test (6MWT) is widely used as an instrument for assessing the functional capacity of cardiac patients. It's a simple, low cost test that better reflects day-to-day activities when compared to other tests. Its use to evaluate the functional capacity of cardiac patients in the in-hospital phase after acute myocardial infarction requires further studies. Objective: To evaluate the safety of the 6MWT performed on the third day after acute myocardial infarction (AMI). Methods: It's a cross-sectional study, to be accomplished in Hospital São Paulo - Federal University of Sao Paulo. Individuals, of both genders, aged 18 years and over, will be assessed on the third day after acute myocardial infarction. The 6MWT will be performed according to the norms of the American Thoracic Society. The distance covered during the 6MWT will be measured as weel as adverse events.

ELIGIBILITY:
Inclusion Criteria:

* AMI patients

Exclusion Criteria:

* Previous history of AMI
* Recurrent or refractory pain
* Presence of neuromuscular diseases
* Acute or chronic lung diseases
* Inability to perform the functional test

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Sequential AMI patients admitted to hospitalization in the third day after myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-08-17 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test to measure functional capacity | Third day after acute myocardial infarction
  By 6MWT assessing the functional capacity after acute myocardial infarction

SECONDARY OUTCOMES:
Angina | Third day after acute myocardial infarction
  To assess the occurrence of angina during the 6MWT
Dyspnea | Third day after acute myocardial infarction
  To assess the occurrence of dyspnea during the 6MWT
Pallor | Third day after acute myocardial infarction
  To assess the occurrence of pallor during the 6MWT
Sweating | Third day after acute myocardial infarction
  To assess the occurrence of sweating during the 6MWT
Cramps | Third day after acute myocardial infarction
  To assess the occurrence of cramps during the 6MWT
Lower limbs fatigue | Third day after acute myocardial infarction
  To assess the occurrence of lower limbs fatigue during the 6MWT
Dizziness | Third day after acute myocardial infarction
  To assess the occurrence of dizziness during the 6MWT
Hospitalization stay | Thirty days after acute myocardial infarction
  Duration of stay in the hospital (in days) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Graciana Santos Martinhão, São Paulo, Brazil